CLINICAL TRIAL: NCT00004497
Title: Phase III Randomized Study of UT-15 in Patients With Primary Pulmonary Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/14287; UTC-FDR001545; UTC-P01-04
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-09

CONDITIONS: Pulmonary Hypertension
Keywords: cardiovascular and respiratory diseases; hypertensive disorder; primary pulmonary hypertension; rare disease
MeSH Terms: conditions — Hypertension, Pulmonary; Respiratory Tract Diseases; Hypertension; Familial Primary Pulmonary Hypertension; Rare Diseases | interventions — treprostinil

INTERVENTIONS:
Drug: UT-15

SUMMARY:
OBJECTIVES:

I. Determine the safety and efficacy of UT-15 in patients with severe symptomatic primary pulmonary hypertension.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified according to center and etiology of disease.

Patients receive conventional oral therapy plus a continuous subcutaneous infusion of either UT-15 or placebo for 12 weeks.

After completing 12 weeks of treatment, patients may continue therapy with open label UT-15. Patients who received placebo cross over to receive UT-15.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of moderate to severe precapillary pulmonary hypertension (New York Heart Association class III/IV) unresponsive to attempted use of chronic oral vasodilators for at least 1 month

Cardiac catheterization at baseline: Pulmonary artery pressure at least 25 mm Hg AND Pulmonary capillary wedge pressure or left ventricular end diastolic pressure no greater than 15 mm Hg AND Pulmonary vascular resistance greater than 3 mm Hg/L/min

Echocardiogram at baseline: Right ventricular hypertrophy or dilation AND Normal left ventricular function AND Absence of mitral valve stenosis

Chest radiograph within prior 3 months Clear lung fields OR Multiple patchy interstitial (not diffuse) lung fields AND At least 1 of the following:

* Right ventricular enlargement
* Prominence of main pulmonary artery
* Enlarged hilar vessels
* Decreased peripheral vessels

No significant parenchymal lung disease within prior 3 months as evidenced by: Total lung capacity no greater than 70% predicted FEV/FVC ratio no greater than 50% Diffuse interstitial fibrosis or alveolitis by high resolution CT if total lung capacity is 70-80% or DLCO less than 60%

No chronic thromboembolic disease with clot proximal to lobar bifurcation

Baseline exercise capacity at least 50 meters walked in six minutes

--Prior/Concurrent Therapy--

Endocrine therapy:

* At least 30 days since prior chronic prostaglandin or prostaglandin analogue therapy (including Flolan IV)
* No concurrent prostaglandins or prostaglandin analogues

Other:

* At least 1 month since prior new type of chronic therapy (e.g., different category of vasodilator, diuretic, digoxin) for pulmonary hypertension, except anticoagulants
* At least 1 week since discontinuation of prior pulmonary hypertension medication, except anticoagulants
* At least 30 days since prior participation in an investigational drug study
* No other concurrent investigational drug
* No concurrent chronic intravenous or inhaled medications (except oxygen)

--Patient Characteristics--

Cardiovascular:

* No portal hypertension
* No left sided heart disease as defined by: Pulmonary capillary wedge pressure or left ventricular end diastolic pressure greater than 15 mm Hg OR LVEF less than 40% by MUGA or angiography OR LV shortening fraction less than 22% by echocardiography OR Symptomatic coronary disease (demonstrable ischemia)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Mentally and physically capable of using an infusion pump
* HIV negative
* No other disease associated with pulmonary hypertension (sickle cell anemia, schistosomiasis)
* No musculoskeletal disorder (arthritis, artificial leg, etc.) or any disease limiting ambulation, or connected to a nonportable machine
* No concurrent physiological condition contraindicating use of UT-15

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-10; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: James Walker Crow, Study Chair — United Therapeutics
Locations (7):
- United States (7):
  - Los Angeles County Harbor-UCLA Medical Center, Torrance, California
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Maryland Medical System, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University College of Physicians and Surgeons, New York, New York
  - United Therapeutics Corporation, Research Triangle Park, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee